CLINICAL TRIAL: NCT05928312
Title: The Efficacy and Safety of Fruquintinib Combined With Chemotherapy as Third-line /Third-line+ Treatment in Advanced Colorectal Cancer: An Open， Single-center Study
Brief Title: Fruquintinib Combined With Chemotherapy as Third-line /Third-line+ Treatment in Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wangxia LV, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C127
Record Dates: First submitted 2023-06-19; First posted 2023-07-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced CRC (Experimental): Patients with Advanced CRC were given Fruquintinib Combine With Chemotherapy.
  Interventions: Drug: Fruquintinib Combined With Chemotherapy

INTERVENTIONS:
Drug: Fruquintinib Combined With Chemotherapy — 1.Security introduction period:
  [1] Safety introduction period (N=6), fruquintinib combined with three-week regimen:
  1. Fruquintinib: Three-week regimen of combined chemotherapy: 4mg/d, orally, once a day, taking the drug for 2 weeks and stopping the drug for 1 week, 3 weeks as a treatment cycle.
  [2] Safety introduction period (N=6), fruquintinib combined 2-week regimen:
  1. Fruquintinib: two-week combination chemotherapy regimen: 4mg/d, orally, once a day, taking the drug for 3 weeks and stopping the drug for 1 week, 4 weeks as a treatment cycle.
  2. Dose expansion phase design(N=60) Cohort 1 (30 patients) : Fruquintinib combined with oxaliplatin. Cohort 2 (30 patients) : Fruquintinib combined with irinotecan .
  Other Names: Fruquintinib oxaliplatin irinotecan

SUMMARY:
To explore the efficacy and safety of fruquintinib combined with chemotherapy as third-line/third-line+ Treatment in advanced metastatic colorectal cancer

DETAILED DESCRIPTION:
Due to the limited efficacy of third-line treatment, the previously effective chemotherapy regimen is a new treatment mode. RE-OPEN, RE-OX and a Korean study confirmed that mCRC patients who had previously been effectively treated with oxaliplatin were retreated with oxaliplatin on the third line to help them achieve OS for 14.5 to 18.5 months. At the same time, a phase III randomized SUNLIGHT study showed good efficacy at the ASCO-GI Congress in 2023. The above studies show that the regimen of antivascular drugs combined with chemotherapy has a tendency to improve the survival of patients with third-line advanced colorectal cancer.

In order to further improve the efficacy of fruquintinib, we conducted a clinical study of fruquintinib combined with chemotherapy to observe the efficacy and safety of Third-line/Third-line+ treatment of advanced colorectal cancer, and to provide a more effective treatment plan for third-line and above treatment for advanced colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent
2. Age ≥18 years old, male or female
3. Advanced metastatic colorectal adenocarcinoma confirmed by histopathology
4. The best efficacy evaluation of first-line chemotherapy (mFOLFOX6, XELOX, or FOLFIRI) in previous patients must be partial response (PR) or above or progression-free survival (PFS) ≥1 year, with a first-line drug withdrawal interval of more than 1 year. Pre-adjuvant/neoadjuvant therapy is allowed. If recurrence or metastasis occurs during or within 6 months after completion of adjuvant/neoadjuvant therapy, adjuvant/neoadjuvant therapy is considered a failure of first-line chemotherapy for advanced disease
5. The patient has failed at least previous second-line treatment，The use of Cetuximab (KRAS and Braf wild type) and bevacizumab in previous anti-tumor regiments is required，Prior treatment with regorafenib or TAS-102 is permitted
6. ECOG status 0-2 points
7. Expected survival ≥12 weeks
8. Have at least one measurable lesion (RECIST version 1.1)
9. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values: Absolute neutrophil count (ANC) ≥1.5×109/L Platelet count ≥80×109 / L Hemoglobin≥80 g/L（<8 g/dL） Serum albumin ≥3g/dL Alanine aminotransferase <2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or <5 × ULN in the presence of liver metastases. Aspartate aminotransferase (AST) <2.5 × ULN if no demonstrable liver metastases or < 5 × ULN in the presence of liver metastases. Total bilirubin (TBL)<1.5 × ULN Creatinine≤ 1.5 × ULN concurrent with creatinine clearance ≤50 mL/min (measured or calculated by the Cockcroft-Gault equation) confirmation of creatinine clearance is only required when creatinine is ≤1.5 × ULN.
10. Fertile male or female patients voluntarily used effective contraceptive methods, such as double barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and within 6 months of the last study dose. All female patients will be considered fertile unless they have undergone natural menopause, artificial menopause, or sterilization (such as hysterectomy, bilateral adnexectomy, or irradiation of radioactive ovaries).
11. Good compliance, cooperate with follow-up.

Exclusion Criteria:

* 1: Patients with known dMMR or MSI-H colorectal cancer who have not previously used anti-PD-1 or PD-L1 inhibitors

  2: Previously received small molecule targeted drug therapy with fuquinitinib

  3: Symptomatic brain or meningeal metastases (except those with brain metastases that have undergone local radiotherapy or surgery for more than 6 months and whose disease control is stable)

  4: Severe infection (such as intravenous infusion of antibiotics, antifungals, or antiviral drugs) within 4 weeks prior to treatment, or unexplained fever > 38.5 ° C during screening/first administration

  5: Have high blood pressure that is not well controlled by antihypertensive medications (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg)

  6: Obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months prior to treatment (bleeding > 30 mL within 3 months, hematemesis, black stool, blood in the stool), hemoptysis (> 5 mL of fresh blood within 4 weeks), etc. Or treatment of arterial venous thrombosis events within the preceding 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism

  7: Long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day) is required

  8: During screening, it was found that the tumor invaded large vascular structures, such as pulmonary artery, superior vena cava or inferior vena cava, etc., and the researchers judged that there was a risk of major bleeding

  9: The patient currently has gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectosed tumors, or other conditions determined by researchers that may cause gastrointestinal bleeding or perforation .Active heart disease, including myocardial infarction, severe/unstable angina, occurs 6 months before treatment. Left ventricular ejection fraction <50% by echocardiography showed poor arrhythmia control.

  10: Patients with other malignant tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) in the past 5 years or at the same time

  11: Known allergy to the investigational drug or any of its excipients

  12: Active or uncontrolled severe infection
  1. Known human immunodeficiency virus (HIV) infection
  2. Known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or >2000 IU/ml) must be excluded for known hepatitis B virus (HBV) carriers
  3. Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis]

  13. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, in which, in the investigator's judgment, there is reason to suspect that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk

  14. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein quantity >1.0g.

  15. Incomplete healing of skin wounds, surgical sites, trauma sites, severe mucosal ulcers or fractures

  16. Stroke events and/or transient cerebral ischemia occurred within 12 months prior to enrollment

  17. The patient has any current disease or condition that affects drug absorption, or the patient is unable to take fuquintinib orally

  18. Women who are pregnant (positive pregnancy test before medication) or breastfeeding

  19. The patients considered by the investigators to be unsuitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2025-06-28 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | up to 12 months
  Usually refers to the highest dose at which a subject's probability of developing DLT does not exceed the probability of target toxicity during the regime-specified DLT observation period.
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib Combine With Immunotherapy and Chemotherapy as second-line therapy to Advanced CRC, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival time | up to 36 months
  OS was calculated from the date of pharmacy to death from any cause.
Assess the anti-tumor activity:DCR | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Wangxia Lv, Study Chair — Zhejiang Cancer Institute & Hospital
Locations (1):
- Zhejiang Cancer Institute & Hospital, Hangzhou, Zhejing, China